CLINICAL TRIAL: NCT06457074
Title: Finerenone for Patients With Primary Aldosteronism (FAIRY): A Multicenter, Randomized Clinical Trial
Brief Title: Finerenone for Patients With Primary Aldosteronism (FAIRY)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qifu Li (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Changzhi Medical College (Other)
Responsible Party: Sponsor-Investigator, Qifu Li, Primary investigator, Chongqing Medical University
Organization: Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAIRY Study
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Primary Aldosteronism
Keywords: Primary aldosteronism; Finerenone; Spironolactone; Antihypertensive effect; Safety
MeSH Terms: conditions — Hyperaldosteronism | interventions — finerenone; Spironolactone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Finerenone (Experimental): Patients divided into Finerenone group need to be treated with finerenone.
  Interventions: Drug: Finerenone Oral Tablet
- Spironolactone (Active Comparator): Patients divided into Spironolactone group need to be treated with spironolactone.
  Interventions: Drug: Spironolactone Oral Tablet

INTERVENTIONS:
Drug: Finerenone Oral Tablet — Eligible patients will be started finerenone at 20mg per day, Dose will be adjusted every four weeks to achieve the targeted blood pressure (the mean office blood pressure <140/90 mmHg).
  Other Names: Finerenone
  Arms: Finerenone
Drug: Spironolactone Oral Tablet — Eligible patients will be started spironolactone at 20mg per day, Dose will be adjusted every four weeks to achieve the targeted blood pressure (the mean office blood pressure <140/90 mmHg).
  Other Names: Spironolactone
  Arms: Spironolactone

SUMMARY:
Using spironolactone as the control, to assess the efficacy and safety of finerenone in patients with primary aldosteronism(PA).

DETAILED DESCRIPTION:
This is a multicenter, randomized study designed to evaluate efficacy and safety of finerenone in patients with PA. PA patients are randomly divided into two groups and treated with finerenone or spironolactone for 12 weeks. Spironolactone will be used as the control, while outcome will be assessed after 12-week treatment. Both drugs will be started at 20mg per day, Dose will be adjusted every four weeks to achieve the targeted blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. . Aged between 18-75, male or female;
2. . With confirmed PA diagnosis (screening positive and at least one confirmatory test is positive); NOTE: Screening positive was defined as plasma aldosterone-to-renin ratio (ARR)

   ≥ 20(pg/ml)/(μIU/ml) or ARR≥30(ng/dL)/(ng/ml/hr). Plasma aldosterone concentration (PAC) post captopril challenge test (CCT) ≥ 110 pg/ml or PAC post seated saline infusion test (SSIT) ≥ 80 pg/ml was considered positive. Note: ARR≥10(pg/ml)/(μIU/ml) or ARR≥15(ng/dL)/(ng/ml/hr) can be considered positive if the patients with hypokalemia (serum potassium < 3.5mmol/L) or adrenal nodules (diameter > 1cm).
3. . Not taking any antihypertensive drugs or on a stable regimen of antihypertensive agents(Limited to alpha-adrenergic receptor blockers and calcium channel blockers.) for more than four weeks before screening;
4. . With a mean seated office SBP≥140 or DBP≥90 mmHg;
5. . Able and willing to give informed consent for participation in the clinical study;

Exclusion Criteria:

1. Has a plan to conduct PA subtype classification(eg. Adrenal vein sampling, PET-CT) in 3 months；
2. Has planned surgery within 3 months;
3. With a mean seated office SBP ≥ 180mmHg or DBP ≥ 110mmHg before randomization; Note: Mean seated BP is defined as the average of 3 seated BP measurements at any single clinical site visit. If the patient did not take their regularly scheduled antihypertensive medications prior to the visit, 1 BP re-test is allowed within 2 days after taking the medications.
4. Night shift workers;
5. Has a body mass index(BMI) ≥30 kg/m2 at screening;
6. Has uncontrolled diabetes with fasting blood glucose(FBG)≥13.3mmol/L at screening;
7. Has uncontrolled chronic diseases;
8. Has known other secondary hypertension (eg, renal artery stenosis, Cushing's syndrome, pheochromocytoma, or aortic coarctation) except subclinical Cushing's syndrome;
9. Has known and documented heart failure (New York Heart Association (NYHA) class III or IV), liver transaminase levels were more than 2 times higher than the upper limit of normal;
10. Has had CABG or other major cardiac surgery (eg, valve replacement), peripheral arterial bypass surgery, or PCI within 6 months before Screening;
11. Has had a stroke, transient ischemic attack, hypertensive encephalopathy, acute coronary syndrome, or hospitalization for heart failure within 6 months before screening;
12. Has poor compliance that can not fully participating in the study;
13. Has hyperkalemia with serum potassium > 5.0mmol/L without potassium supplementation;
14. Has a history of uncontrolled malignant tumor;
15. Has more than 20mmHg difference of seated office SBP in both arms;
16. Is not willing or not able to stop taking sex hormones, glucocorticoids, non-steroidal anti-inflammatory drugs, cyclosporine, tacrolimus, or antidepressants;
17. Is pregnant, breastfeeding, or planning to become pregnant during the study;
18. Complicated with severe mental illness;
19. Has had prior solid organ transplant and/or cell transplants;
20. Has a history of allergy to Finerenone or spironolactone;
21. Has typical consumption of ≥15 alcoholic drinks weekly. Note: 1 drink of alcohol is equivalent to 360ml beer, 45ml spirits, or 150ml wine;
22. Has participated in another clinical study involving any investigational drug within 30 days prior to screening；
23. Female of childbearing potential refuses to use non-hormonal contraception methods during the study period;
24. Refuse to stop eating grapefruit or grapefruit juice during treatment with Finerenone;
25. Other situations that the investigator assesses the subject as unable to complete the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 24-hour SBP | 12 weeks
  Change from baseline in 24-hour systolic blood pressure (SBP) assessed by 24-hour ambulatory blood pressure monitoring compared to spironolactone after 12 weeks of finerenone therapy in patients with PA.

SECONDARY OUTCOMES:
Change from baseline in 24-hour DBP | 12 weeks
  Change from baseline in 24-hour diastolic blood pressure (DBP) assessed by 24-hour ambulatory blood pressure monitoring compared to spironolactone after 12 weeks of finerenone therapy in patients with PA.
Change from baseline in daytime SBP | 12 weeks
  Change from baseline in daytime systolic blood pressure (SBP) assessed by 24-hour ambulatory blood pressure monitoring compared to spironolactone after 12 weeks of finerenone therapy in patients with PA.
Change from baseline in daytime DBP | 12 weeks
  Change from baseline in daytime diastolic blood pressure (DBP) assessed by 24-hour ambulatory blood pressure monitoring compared to spironolactone after 12 weeks of finerenone therapy in patients with PA.
Change from baseline in nighttime SBP | 12 weeks
  Change from baseline in nighttime systolic blood pressure (SBP) assessed by 24-hour ambulatory blood pressure monitoring compared to spironolactone after 12 weeks of finerenone therapy in patients with PA.
Change from baseline in nighttime DBP | 12 weeks
  Change from baseline in nighttime diastolic blood pressure (DBP) assessed by 24-hour ambulatory blood pressure monitoring compared to spironolactone after 12 weeks of finerenone therapy in patients with PA.
Blood pressure control rate at the end of the study | 12 weeks
  Blood pressure control rate was defined as the number of patients with blood pressure controlled (with mean seated office BP<140/90mmHg at the end of the study)/ total number of patients in each group × 100%.
Serum potassium | 12 weeks
  Change from baseline in Serum potassium, Blood was drawn to measure potassium.
Hypokalemia control rate at the end of the study | 12 weeks
  Hypokalemia control rate was defined as the number of hypokalemic patients with serum potassium>3.5mmol/l at the end of the study/number of hypokalemic patients at baseline× 100%.
Plasma renin concentration | 12 weeks
  Change from baseline in plasma renin concentration,Blood was drawn to measure renin.

OTHER OUTCOMES:
Proportion of subjects with AEs | 12 weeks
  Adverse events(AEs) defined as any untoward medical occurrence in a clinical investigation that occurs to a patient administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment.
Proportion of subjects with SAEs and AEs leading to discontinuation of treatment with study drug | 12 weeks
  Serious adverse events(SAEs) results in any of the following outcomes:Death;A life-threatening AE;Requires hospitalization or prolongation of existing hospitalizations;A persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions.
Change in eGFR from baseline. | 12 weeks
  Blood was drawn to measure eGFR（mL/min/1.73m2）
Change from baseline in urinary albumin-to-creatinine ratio(UACR) | 12 weeks
  Urine will be collected to measure UACR
Change from baseline in urinary Change in the UACR from baseline>30(mg/g Cr). | 12 weeks
  Urine will be collected to measure UACR

CONTACTS AND LOCATIONS:
Overall Officials: Shumin Yang, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- the first affiliated hospital of Chongqing medical university, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rehan M, Raizman JE, Cavalier E, Don-Wauchope AC, Holmes DT. Laboratory challenges in primary aldosteronism screening and diagnosis. Clin Biochem. 2015 Apr;48(6):377-87. doi: 10.1016/j.clinbiochem.2015.01.003. Epub 2015 Jan 22. PMID 25619896
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Menard J. The 45-year story of the development of an anti-aldosterone more specific than spironolactone. Mol Cell Endocrinol. 2004 Mar 31;217(1-2):45-52. doi: 10.1016/j.mce.2003.10.008. PMID 15134800
- [Background] Vilela LAP, Almeida MQ. Diagnosis and management of primary aldosteronism. Arch Endocrinol Metab. 2017 May-Jun;61(3):305-312. doi: 10.1590/2359-3997000000274. PMID 28699986
- [Background] Pitt B, Kober L, Ponikowski P, Gheorghiade M, Filippatos G, Krum H, Nowack C, Kolkhof P, Kim SY, Zannad F. Safety and tolerability of the novel non-steroidal mineralocorticoid receptor antagonist BAY 94-8862 in patients with chronic heart failure and mild or moderate chronic kidney disease: a randomized, double-blind trial. Eur Heart J. 2013 Aug;34(31):2453-63. doi: 10.1093/eurheartj/eht187. Epub 2013 May 27. PMID 23713082
- [Background] Agarwal R, Ruilope LM, Ruiz-Hurtado G, Haller H, Schmieder RE, Anker SD, Filippatos G, Pitt B, Rossing P, Lambelet M, Nowack C, Kolkhof P, Joseph A, Bakris GL. Effect of finerenone on ambulatory blood pressure in chronic kidney disease in type 2 diabetes. J Hypertens. 2023 Feb 1;41(2):295-302. doi: 10.1097/HJH.0000000000003330. Epub 2022 Dec 8. PMID 36583355
- [Background] Agarwal R, Pitt B, Palmer BF, Kovesdy CP, Burgess E, Filippatos G, Malyszko J, Ruilope LM, Rossignol P, Rossing P, Pecoits-Filho R, Anker SD, Joseph A, Lawatscheck R, Wilson D, Gebel M, Bakris GL. A comparative post hoc analysis of finerenone and spironolactone in resistant hypertension in moderate-to-advanced chronic kidney disease. Clin Kidney J. 2022 Oct 30;16(2):293-302. doi: 10.1093/ckj/sfac234. eCollection 2023 Feb. PMID 36864892
- [Background] Filippatos G, Anker SD, Agarwal R, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Schloemer P, Tornus I, Joseph A, Bakris GL; FIDELIO-DKD Investigators. Finerenone and Cardiovascular Outcomes in Patients With Chronic Kidney Disease and Type 2 Diabetes. Circulation. 2021 Feb 9;143(6):540-552. doi: 10.1161/CIRCULATIONAHA.120.051898. Epub 2020 Nov 16. PMID 33198491
- [Background] Bakris GL, Agarwal R, Chan JC, Cooper ME, Gansevoort RT, Haller H, Remuzzi G, Rossing P, Schmieder RE, Nowack C, Kolkhof P, Joseph A, Pieper A, Kimmeskamp-Kirschbaum N, Ruilope LM; Mineralocorticoid Receptor Antagonist Tolerability Study-Diabetic Nephropathy (ARTS-DN) Study Group. Effect of Finerenone on Albuminuria in Patients With Diabetic Nephropathy: A Randomized Clinical Trial. JAMA. 2015 Sep 1;314(9):884-94. doi: 10.1001/jama.2015.10081. PMID 26325557
- [Background] Song Y, Yang S, He W, Hu J, Cheng Q, Wang Y, Luo T, Ma L, Zhen Q, Zhang S, Mei M, Wang Z, Qing H, Bruemmer D, Peng B, Li Q; Chongqing Primary Aldosteronism Study (CONPASS) Groupdagger. Confirmatory Tests for the Diagnosis of Primary Aldosteronism: A Prospective Diagnostic Accuracy Study. Hypertension. 2018 Jan;71(1):118-124. doi: 10.1161/HYPERTENSIONAHA.117.10197. Epub 2017 Nov 20. PMID 29158354
- [Background] Thuzar M, Young K, Ahmed AH, Ward G, Wolley M, Guo Z, Gordon RD, McWhinney BC, Ungerer JP, Stowasser M. Diagnosis of Primary Aldosteronism by Seated Saline Suppression Test-Variability Between Immunoassay and HPLC-MS/MS. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz150. doi: 10.1210/clinem/dgz150. PMID 31676899
- [Background] Mulatero P, Monticone S, Deinum J, Amar L, Prejbisz A, Zennaro MC, Beuschlein F, Rossi GP, Nishikawa T, Morganti A, Seccia TM, Lin YH, Fallo F, Widimsky J. Genetics, prevalence, screening and confirmation of primary aldosteronism: a position statement and consensus of the Working Group on Endocrine Hypertension of The European Society of Hypertension. J Hypertens. 2020 Oct;38(10):1919-1928. doi: 10.1097/HJH.0000000000002510. PMID 32890264
- [Background] Muntner P, Shimbo D, Carey RM, Charleston JB, Gaillard T, Misra S, Myers MG, Ogedegbe G, Schwartz JE, Townsend RR, Urbina EM, Viera AJ, White WB, Wright JT Jr. Measurement of Blood Pressure in Humans: A Scientific Statement From the American Heart Association. Hypertension. 2019 May;73(5):e35-e66. doi: 10.1161/HYP.0000000000000087. PMID 30827125
- [Background] Bakris GL, Agarwal R, Anker SD, Pitt B, Ruilope LM, Rossing P, Kolkhof P, Nowack C, Schloemer P, Joseph A, Filippatos G; FIDELIO-DKD Investigators. Effect of Finerenone on Chronic Kidney Disease Outcomes in Type 2 Diabetes. N Engl J Med. 2020 Dec 3;383(23):2219-2229. doi: 10.1056/NEJMoa2025845. Epub 2020 Oct 23. PMID 33264825
- [Background] Mancia G, Kreutz R, Brunstrom M, Burnier M, Grassi G, Januszewicz A, Muiesan ML, Tsioufis K, Agabiti-Rosei E, Algharably EAE, Azizi M, Benetos A, Borghi C, Hitij JB, Cifkova R, Coca A, Cornelissen V, Cruickshank JK, Cunha PG, Danser AHJ, Pinho RM, Delles C, Dominiczak AF, Dorobantu M, Doumas M, Fernandez-Alfonso MS, Halimi JM, Jarai Z, Jelakovic B, Jordan J, Kuznetsova T, Laurent S, Lovic D, Lurbe E, Mahfoud F, Manolis A, Miglinas M, Narkiewicz K, Niiranen T, Palatini P, Parati G, Pathak A, Persu A, Polonia J, Redon J, Sarafidis P, Schmieder R, Spronck B, Stabouli S, Stergiou G, Taddei S, Thomopoulos C, Tomaszewski M, Van de Borne P, Wanner C, Weber T, Williams B, Zhang ZY, Kjeldsen SE. 2023 ESH Guidelines for the management of arterial hypertension The Task Force for the management of arterial hypertension of the European Society of Hypertension: Endorsed by the International Society of Hypertension (ISH) and the European Renal Association (ERA). J Hypertens. 2023 Dec 1;41(12):1874-2071. doi: 10.1097/HJH.0000000000003480. Epub 2023 Sep 26. PMID 37345492

DOCUMENTS (1):
  • Study Protocol (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT06457074/Prot_001.pdf